CLINICAL TRIAL: NCT06166160
Title: Clinical Performance of a Flowable Bulk Fill Composite Versus a Highly Viscous Glass-ionomer Cement in Restoring Class II Cavities of Primary Molars: A Randomized Clinical Trial
Brief Title: Clinical Performance of a Flowable Bulk Fill Composite Versus a Highly Viscous Glass-ionomer Cement in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marina F Fahmy, MD, Assistant lecturer of pdiateric dentistry and dental public health ,faculty of dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PED22-3D
Record Dates: First submitted 2023-11-20; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Management of Dental Caries of Primary Molars
Keywords: bulk-fill flowable composite , high viscous GIC ,

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDR FLOW + bulk fill flowable (Experimental): in class II cavities of primary molars
  Interventions: Other: Bulk fill flowable composite SDR Dentsply sirona
- high-viscosity glass ionomer cement (EQUIA Forte) (Active Comparator): in class II cavities of primary molars
  Interventions: Other: Bulk fill flowable composite SDR Dentsply sirona

INTERVENTIONS:
Other: Bulk fill flowable composite SDR Dentsply sirona — caries removal in class II cavities of primary molars and application of experminted restorations
  Other Names: high viscosity glass ionomer cement (EQUIA Forte HT) GC

SUMMARY:
the study was conducted to compare and evaluate the clinical performance of EQUIA Forte and SDR® flow+ in class II cavities in primary molar

DETAILED DESCRIPTION:
Initial intra-oral periapical bitewing radiographs of the teeth to be treated were taken before the procedure. After obtaining partial isolation using cotton rolls and saliva ejector, caries excavation and removal of undermined enamel will be done using high-speed diamond burs with water cooling and hand instruments. After finishing the cavity, a matrix band will be placed with the interproximal wedge. The prepared cavities will be restored using Equia Forte or flowable bulk-fill composite resin according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

1. 4 to 8 years old medically free children.
2. Cooperative children are classified as class 3 or 4 based on Frankel et al. classification.
3. Children who had at least one active dentinal carious lesion on the proximal surface of primary molars

Exclusion Criteria:

1. Refusal of the parents to sign the informed consent
2. Presence of deep bite or any pictures of malocclusion and parafunctional habits.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical performance | one-year
  The difference in the clinical performance flowable bulk fill composite SDR® flow+ and and high viscous glass-ionomer cement(EQUIA Forte) In Class II cavities in primary molars using FDI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marina F Fahmy, ass.lecturer, Principal Investigator — assistant lecturer of pediatric dentistry ,faculty of dentistry ASU
Locations (2):
- Egypt (2):
  - Faculty of dentistry .Ain shams university, Cairo
  - Marina Fakhry Fahmy, Cairo

IPD SHARING:
Plan to Share IPD: No
study protocol